CLINICAL TRIAL: NCT04902118
Title: Burnout Determinants Among Pediatric Psychiatry Workers During COVID-19 Epidemic in Occitanie Region in France
Brief Title: Burnout Determinants Among Pediatric Psychiatry Workers During COVID-19 Crisis
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0305
Record Dates: First submitted 2021-05-25; First posted 2021-05-26 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Burnout
Keywords: Burnout status
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Burnout among health workers is at core of our current preoccupations because of the health crisis we're going trough. Indeed, COVID-19 epidemic had terrible consequences not only on global mental health both in adults and children, but also on Health workers mental health. The investigators chose to consider Pediatric Psychiatry workers because of their particular position in this crisis.

The aim of the study is to point out burnout determining factors among Pediatric Psychiatry workers in Occitanie during COVID-19 crisis, by the use of an online questionnaire including the Copenhagen Burnout Inventory.

ELIGIBILITY:
Inclusion criteria:

- Medical doctors, interns, Paramedics (nurse, assistant nurse), Psychologists, Caseworkers working > 50% in a structure medico socio sanitaire

Exclusion criteria:

- Other persons working in a in a structure medico socio sanitaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical and paramedical workers in the field of Pediatric Psychiatry in the Occitanie region
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Copenhagen Burnout Inventory | 1 day
  Copenhagen Burnout Inventory, comprising two subscales assessing general and patients-related burnout.

SECONDARY OUTCOMES:
Epidemic attribuable stress proportion | 1 day
  Declarative quantitative assessment of COVID-19 epidemic attribuable stress proportion

CONTACTS AND LOCATIONS:
Overall Officials: Diane Purper-Ouakil, M.D., Ph. D., Principal Investigator — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC